CLINICAL TRIAL: NCT04053439
Title: A Single Centre Cohort Study to Determine if Clonal Hematopoieses of Indeterminate Potential (CHIP) is a Risk Factor for Chemotherapy-Related Complications in Lymphoma Patients >= 60 Receiving Cytotoxic Chemotherapy
Brief Title: Clonal Hematopoiesis is a Risk Factor for Chemotherapy-Related Complications
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: The Leukemia and Lymphoma Society (Other); Queen's University (Other)
Responsible Party: Sponsor
Other Study IDs: CHIP Lymphoma
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma; Chemotherapeutic Toxicity
Keywords: Clonal Hematopoiesis of Indeterminate Significance; Chemotherapy; Lymphoma; Chemotherapy complications
MeSH Terms: conditions — Lymphoma | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A peripheral blood ethylenediaminetetraacetic acid (EDTA) tube will be used to obtain blood for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lymphoma patients >=60 receiving cytotoxic chemotherapy: Lymphoma patients >=60 receiving cytotoxic chemotherapy who have consented to DNA extraction and analysis for CHIP.
  Interventions: Other: Blood test for determination of CHIP

INTERVENTIONS:
Other: Blood test for determination of CHIP — Patients will have one additional blood draw to be sent for DNA extraction and sequencing for CHIP.

SUMMARY:
'CHIP' stands for Clonal Hematopoiesis of Indeterminate Significance, which are mutations in bone marrow stem cells that give that population of cells a survival or 'clonal' advantage for growth. This study investigates whether CHIP in lymphoma patients aged 60 years and older is a risk factor for chemotherapy-related complications like low blood counts, infections, cardiac events, hospitalizations, dose delays and dose reductions, and failure to recover normal blood counts after chemotherapy finishes.

DETAILED DESCRIPTION:
'CHIP' stands for Clonal Hematopoiesis of Indeterminate Significance (1-4). Up to 20% of individuals in the general population acquire mutations in their bone marrow stem cells as they age that give that population of cells a survival or 'clonal' advantage for growth. The frequency of CHIP may be higher in patients with other cancers. CHIP increases with age, and has been shown to be a risk factor associated with cardiovascular disease and a tendency to the development of bone marrow cancers at a rate of 1% per year (1,2,5). CHIP is also associated with the development of bone marrow cancers that occur after chemotherapy. The investigators want to investigate whether CHIP is also a risk factor for chemotherapy-related complications like low blood counts, infections, cardiac events, hospitalizations, dose delays and dose reductions. They are also interested in determining if CHIP may explain why some patients do not recover normal blood counts after chemotherapy finishes.

The results from this study may help physicians better understand why some people have difficulty with chemotherapy (in the short and long-term) while others do not. Screening for CHIP in older patients may become a recommended standard that allows physicians to tailor anti-cancer treatment to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a lymphoma (ex: diffuse large B cell lymphoma (DLBCL), follicular lymphoma, marginal zone lymphoma, small lymphocytic lymphoma/chronic lymphocytic leukemia, Hodgkin's lymphoma, peripheral T cell lymphoma, anaplastic large cell lymphoma, angioimmunoblastic lymphoma, hairy cell leukemia, Waldenstrom's macroglobulinemia, anaplastic large cell lymphoma, small lymphocytic lymphoma/chronic lymphocytic leukemia, and mantle cell lymphoma).
* Commencing first or second-line cytotoxic chemotherapy for lymphoma with or without rituximab [ex: cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP), cyclophosphamide, vincristine and prednisone (CVP), Fludarabine, fludarabine cyclophosphamide (FC), Bendamustine, cisplatin, cytarabine, dexamethasone (DHAP), etoposide, cytarabine, cisplatin, prednisone (ESHAP), gemcitabine, cisplatin and dexamethasone (GDP), Cladribine, Cyclophosphamide, Epirubicin, Vincristine, Prednisone (CEOP), dose-adjusted Dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (DA-EPOCH)]

Exclusion Criteria:

* Pre-existing diagnosis of myeloid neoplasm
* Circulating lymphocyte count > 10 x 109/L
* Significant uncontrolled renal or hepatic impairment [>1.5 x upper limit of normal (ULN) bilirubin, >1.5 x ULN Alanine aminotransferase (ALT), >1.5 x ULN creatinine]
* HIV
* Active infection

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Elderly patients (>= 60 years old) being treated at a tertiary cancer centre in Toronto, ON.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Determine if CHIP is an independent risk factor for chemotherapy-induced complications. | Up to 24 weeks
  Complications during chemotherapy defined as any or all of the following: febrile neutropenia, new grades 3-4 anemia, thrombocytopenia and neutropenia immediately (day -1 or 0) preceding next cycle of chemotherapy, secondary dose reductions or dose delays due to myelosuppression or toxicity, cardiovascular toxicity (arrhythmias, congestive heart failure, symptomatic coronary disease), secondary granulocyte colony-stimulating factor (GCSF) use due to neutropenia, inability to complete all scheduled cycles due to chemotherapy related complications, dose delays that exceed 7 days.
Emerging dysmyelopoiesis after chemotherapy | Up to 12 months after completion of chemotherapy
  The number of patients with and without CHIP who, following at 6 and 12 months post chemotherapy have:
  1. Hemoglobin, white blood cell (WBC) or platelet (PLT) count that does not recover to normal pre-chemotherapy levels
  2. Persistant macrocytosis defined as mean cell volume (MCV) > 96 fl
  3. Persistant anisocytosis defined as red cell distribution width (RDW) > 14.5%

SECONDARY OUTCOMES:
Expansion of clonal hematopoietic stem cells | Up to 5 years after completion of chemotherapy
  Expansion of clonal hematopoietic stem cells over time measured using next generation sequencing of 40 myeloid genes in patients with CHIP at baseline defined by variant allele frequency (VAF) that increases by 10% of more or the emergence of new clones
Development of therapy-related myeloid neoplasm | Up to 5 years after completion of chemotherapy
  Therapy-related myeloid neoplasm defined as any of myelodysplastic syndrome (MDS), acute myeloid leukemia (AML), myeloproliferative neoplasm (MPN), MDS/MPN diagnosed by bone marrow exam
Overall survival | Up to 5 years after completion of chemotherapy
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Rena Buckstein, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre; Hubert Tsui, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Michael Rauh, MD, Principal Investigator — Queen's University
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaiswal S, Fontanillas P, Flannick J, Manning A, Grauman PV, Mar BG, Lindsley RC, Mermel CH, Burtt N, Chavez A, Higgins JM, Moltchanov V, Kuo FC, Kluk MJ, Henderson B, Kinnunen L, Koistinen HA, Ladenvall C, Getz G, Correa A, Banahan BF, Gabriel S, Kathiresan S, Stringham HM, McCarthy MI, Boehnke M, Tuomilehto J, Haiman C, Groop L, Atzmon G, Wilson JG, Neuberg D, Altshuler D, Ebert BL. Age-related clonal hematopoiesis associated with adverse outcomes. N Engl J Med. 2014 Dec 25;371(26):2488-98. doi: 10.1056/NEJMoa1408617. Epub 2014 Nov 26. PMID 25426837
- [Background] Genovese G, Kahler AK, Handsaker RE, Lindberg J, Rose SA, Bakhoum SF, Chambert K, Mick E, Neale BM, Fromer M, Purcell SM, Svantesson O, Landen M, Hoglund M, Lehmann S, Gabriel SB, Moran JL, Lander ES, Sullivan PF, Sklar P, Gronberg H, Hultman CM, McCarroll SA. Clonal hematopoiesis and blood-cancer risk inferred from blood DNA sequence. N Engl J Med. 2014 Dec 25;371(26):2477-87. doi: 10.1056/NEJMoa1409405. Epub 2014 Nov 26. PMID 25426838
- [Background] McKerrell T, Park N, Moreno T, Grove CS, Ponstingl H, Stephens J; Understanding Society Scientific Group; Crawley C, Craig J, Scott MA, Hodkinson C, Baxter J, Rad R, Forsyth DR, Quail MA, Zeggini E, Ouwehand W, Varela I, Vassiliou GS. Leukemia-associated somatic mutations drive distinct patterns of age-related clonal hemopoiesis. Cell Rep. 2015 Mar 3;10(8):1239-45. doi: 10.1016/j.celrep.2015.02.005. Epub 2015 Feb 26. PMID 25732814
- [Background] Xie M, Lu C, Wang J, McLellan MD, Johnson KJ, Wendl MC, McMichael JF, Schmidt HK, Yellapantula V, Miller CA, Ozenberger BA, Welch JS, Link DC, Walter MJ, Mardis ER, Dipersio JF, Chen F, Wilson RK, Ley TJ, Ding L. Age-related mutations associated with clonal hematopoietic expansion and malignancies. Nat Med. 2014 Dec;20(12):1472-8. doi: 10.1038/nm.3733. Epub 2014 Oct 19. PMID 25326804
- [Background] Steensma DP, Bejar R, Jaiswal S, Lindsley RC, Sekeres MA, Hasserjian RP, Ebert BL. Clonal hematopoiesis of indeterminate potential and its distinction from myelodysplastic syndromes. Blood. 2015 Jul 2;126(1):9-16. doi: 10.1182/blood-2015-03-631747. Epub 2015 Apr 30. PMID 25931582